CLINICAL TRIAL: NCT03723434
Title: Physiology of Interregional Connectivity in the Human Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Tommi Raij, Research Scientist, Brain Stimulation Director, Shirley Ryan AbilityLab
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU00204239
Record Dates: First submitted 2018-10-22; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Healthy; Stroke; Traumatic Brain Injury; Multiple Sclerosis
Keywords: Human; Brain; Connectivity; Stroke; Traumatic brain injury; Multiple sclerosis; Transcranial magnetic stimulation; Paired associative stimulation; Electroencephalography; Magnetic resonance imaging
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: PAS will be applied to two cortical targets at different asynchronies to modulate connectivity. PAS may selectively increase or decrease effective connectivity depending on the asynchrony. Negative asynchronies are expected to decrease effective connectivity, whereas positive asynchronies to increase it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Participants (Active Comparator): Healthy participants without disorders or medications influencing brain function will be scanned with MRI and undergo single-pulse TMS and PAS during several visits, each with a different asynchrony, while EEG and MEPs are recorded.
  Interventions: Device: Single-pulse transcranial magnetic stimulation (spTMS); Device: Paired associative stimulation (PAS); Device: Repetitive transcranial magnetic stimulation (rTMS)
- Patients (Experimental): Participants with stroke, traumatic brain injury (TBI), or multiple sclerosis (MS) will be scanned with MRI and undergo single-pulse TMS and paired associative stimulation during several visits while EEG is recorded.
  Interventions: Device: Single-pulse transcranial magnetic stimulation (spTMS); Device: Paired associative stimulation (PAS)

INTERVENTIONS:
Device: Single-pulse transcranial magnetic stimulation (spTMS) — Single-pulse TMS (spTMS) will be delivered with a TMS stimulator (MagPro X100 w/ MagOption, MagVenture, Farum, Denmark) and a figure-of-eight TMS coil. 80 spTMS will be repeated at 0.2 Hz. An MRI-based TMS navigation system will be used to navigate the TMS coil (Localite, St Augustin, Germany).
Device: Paired associative stimulation (PAS) — Paired associative stimulation (PAS) will be applied with two TMS stimulators (MagPro X100 w/ MagOption, MagVenture, Farum, Denmark) and two TMS coils. The pulses from each stimulator/coil will be repeated at 0.2 Hz, duration of run 15 minutes (180 pulses for each stimulator/coil). In different sessions, we will deliver PAS with different asynchrony values to examine their effects on effective connectivity. Coils will be navigated using an MRI-based TMS navigation system (Localite, St Augustin, Germany).
Device: Repetitive transcranial magnetic stimulation (rTMS) — Repetitive TMS (rTMS) will be applied at 1 and 20 Hz with a TMS stimulator (MagPro X100 w/ MagOption, MagVenture, Farum, Denmark) and a figure-of-eight TMS coil. 300 rTMS pulses will be delivered during 1 and 20 Hz stimulation. An MRI-based TMS navigation system will be used to navigate the TMS coil (Localite, St Augustin, Germany).
  Arms: Healthy Participants

SUMMARY:
The purpose of this study is to understand the physiology of connectivity between cortical regions in the human brain in healthy participants and in patients with white matter lesions. Specifically, the investigators will examine the effects of paired associative stimulation (PAS) which consists in delivering brief (< 1 ms) current pulses separated by a short millisecond-level time interval ("asynchrony") to two cortical areas. The used techniques are all non-invasive and considered safe in humans: transcranial magnetic stimulation (TMS), electroencephalography (EEG), magnetic resonance imaging (MRI), and functional MRI (fMRI). Based on prior literature in animals and human studies, it is hypothesized that PAS may increase or decrease effective connectivity between the stimulated areas depending on the asynchrony value. The main outcome measure is source-resolved EEG responses evoked by single-pulse TMS; this is a more direct measure of neuronal changes occurring at the targeted cortical area than motor evoked potentials (MEPs) or sensor-level EEG responses used in previous studies.

DETAILED DESCRIPTION:
This study consists of two experiments.

In Experiment A, healthy participants without disorders or medications influencing brain function (N=24) will be recruited. A range of negative and positive asynchronies (from minus 50 to + 50 ms) will be tested. To allow comparison with prior studies that used MEPs as outcome measures, in 12 participants the primary motor cortex in the left and right hemisphere will be targeted. In another 12 participants, two cortical areas within the same hemisphere will be stimulated.

In Experiment B, participants with stroke, traumatic brain injury (TBI), or multiple sclerosis (MS) (total maximum N across all such participants is 52) will be recruited. These participants are required to have one or more subcortical white matter lesions, which would be expected to result in cortico-cortical disconnections. Here, the investigators will only test PAS with positive asynchronies, with the goal of testing if the findings observed in healthy participants are similar in participants with white matter lesions. It will also be examined if the PAS-induced connectivity changes persist beyond the stimulation sessions if PAS is given repeatedly over several days. PAS will be applied to two cortical targets that have been disconnected from each other. The rationale for including more than one disorder in Experiment B is that the disconnections are in all cases caused by white matter lesions and the results may therefore be similar. To detect possible differences between disorders, the data from the three groups will also be analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Healthy Participants:

* Age from 18 to 85 years
* Right-handed
* Normal hearing and (corrected) vision
* Able to understand and give informed consent
* English speaker

Inclusion Criteria for Patients:

* Age from 18 to 85 years
* Stroke (ischemic subcortical, intermediate level, chronic phase 3 weeks or more from lesion)
* TBI (closed-skull, intermediate level, chronic phase 3 weeks or more from lesion)
* MS (white matter subcortical lesion)
* Clinical and radiological evidence supporting the above diagnoses
* One or more behavioral symptoms possibly linked to the white matter lesion(s)
* Stable medical condition
* English speaker

Exclusion Criteria:

Exclusion Criteria for Healthy Participants:

* Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
* Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
* Surgical clips in the head or previous neurosurgery
* Any magnetic particles in the body
* Cochlear implants
* Prosthetic heart valves
* Epilepsy or any other type of seizure history
* Any neurological diagnoses or medications influencing brain function
* History of significant head trauma (i.e., extended loss of consciousness, neurological sequelae)
* Known structural brain lesion
* Significant other disease (heart disease, malignant tumors, mental disorders)
* Significant claustrophobia; Ménière's disease
* Pregnancy (ruled out by urine ß-HCG if answers to screening questions suggest that pregnancy is possible), breast feeding
* Non prescribed drug use
* Failure to perform the behavioral tasks or neuropsychological evaluation tests
* Prisoners

Exclusion Criteria for Patients:

* Same as above, excluding the requirement of no structural brain lesion, and medications influencing brain function are allowed
* Patients with cortical lesions or CSF-filled cysts/cavities near the TMS sites
* MS patients with acute exacerbation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2017-05-31 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Changes in EEG effective connectivity | Experiment A: Within-session (before versus after PAS at 1 and 60 minutes). Experiment B: Within-session (before versus after PAS at 1 and 60 minutes). Across-sessions (persistence of changes up to 1 month after last PAS session).
  EEG will be recorded with a 64-channel whole-head TMS-compatible device (NeurOne, Bittium, Kuopio, Finland). Data will be collected before (Pre-PAS) and at 1 minute (Post-PAS T1) and at 60 minutes (Post-PAS T60) after PAS. To record spTMS-evoked EEG responses the investigators will deliver 80 single TMS pulses to the two areas receiving PAS, one target after the other in separate runs. Effective connectivity will be measured by comparing the source-resolved EEG evoked response waveforms before (Pre-PAS) and at 1 (Post-PAS T1) and at 60 minutes after PAS (Post-PAS T60).
Changes in resting-state EEG coherence | Experiment A: Within-session (before versus after PAS at 1 and 60 minutes). Experiment B: Within-session (before versus after PAS at 1 and 60 minutes). Across-sessions (persistence of changes up to 1 month after last PAS session).
  Resting-state EEG will be recorded with a 64-channel whole-head device (NeurOne, Bittium, Kuopio, Finland). Data will be collected before (Pre-PAS) and at 1 minute (Post-PAS T1) and at 60 minutes (Post-PAS T60) after PAS. Resting-state EEG coherence will be computed in the source space for the two areas receiving PAS from 1 to 100 Hz.

SECONDARY OUTCOMES:
Motor evoked potentials (MEPs) | Experiment A: Within-session (before versus after PAS at 1 and 60 minutes). Experiment B: Done only in patients where the M1 was targeted with PAS.
  To assess the effects of PAS in participants where the primary motor cortex (M1) was targeted, spTMS will be administered to the M1 at 110% of resting motor threshold (rMT) while MEPs are recorded from the contralateral hand (NeurOne, Bittium, Kuopio, Finland). The MEPs will be recorded before (Pre-PAS), at 1 minute (Post-PAS T1) and at 60 minutes (Post-PAS T60) after PAS.
MRI functional connectivity | Experiment A: Baseline. Experiment B: Baseline to 1 month after the last PAS session.
  Functional connectivity will be assessed with resting-state MRI (rs-MRI).
MRI structural connectivity | Experiment A: Baseline. Experiment B: Baseline to 1 month after the last PAS session.
  Structural connectivity will be assessed with diffusion tensor imaging (DTI).

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Raij, MD, PhD, Principal Investigator — Shirley Ryan AbilityLab 355 East Erie St, Chicago, IL Department of Physical Medicine and Rehabilitation, Feinberg School of Medicine, Northwestern University, Chicago, IL
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States